CLINICAL TRIAL: NCT02972658
Title: A Randomized, Double-Blind, Delayed-Start Study of LY3314814 (AZD3293) in Early Alzheimer's Disease Dementia (Extension of Study AZES, The AMARANTH Study)
Brief Title: A Study of Lanabecestat (LY3314814) in Early Alzheimer's Disease Dementia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: As the feeder study (AZES) was stopped for futility after an independent assessment, this trial was also stopped.
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16557; I8D-MC-AZFD (Other: Eli Lilly and Company); 2016-003440-36 (EudraCT Number)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Dementia; Brain Diseases; Neurodegenerative Diseases; Central Nervous System Diseases; Nervous System Diseases; Mental Disorders; Delirium, Dementia, Amnestic, Cognitive Disorders; Tauopathies; Memory; Amyloid
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Neurodegenerative Diseases; Central Nervous System Diseases; Nervous System Diseases; Mental Disorders; Neurocognitive Disorders; Tauopathies | interventions — lanabecestat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AZES Lanabecestat 20 milligrams (mg)/AZFD Lanabecestat 20 mg (Experimental): Participants who received Lanabecestat 20 mg in the feeder study (AZES) were randomized to receive Lanabecestat 20 mg.
  Interventions: Drug: Lanabecestat
- AZES Lanabecestat 50 mg/AZFD Lanabecestat 50 mg (Experimental): Participants who received Lanabecestat 50 mg in the feeder study (AZES) were randomized to receive Lanabecestat 50 mg.
  Interventions: Drug: Lanabecestat
- AZES Placebo/AZFD Lanabecestat 20 mg (Experimental): Participants who received placebo in the feeder study (AZES) were randomized to receive Lanabecestat 20 mg.
  Interventions: Drug: Lanabecestat
- AZES Placebo/AZFD Lanabecestat 50 mg (Experimental): Participants who received placebo in the feeder study (AZES) were randomized to receive Lanabecestat 50 mg.
  Interventions: Drug: Lanabecestat

INTERVENTIONS:
Drug: Lanabecestat — Administered orally
  Other Names: LY3314814; AZD3293

SUMMARY:
This study is an extension of study I8D-MC-AZES (NCT02245737), the AMARANTH study. The purpose of this study is to evaluate the effectiveness of the study drug lanabecestat in participants with early Alzheimer's disease dementia at the time of entry into study I8D-MC-AZES.

DETAILED DESCRIPTION:
Study AZFD was designed to be integrated with 104-week study AZES to form a Delayed-Start study (Study AZES-FD). Study AZES-FD was to be used to test the hypothesis that participants originally randomized to receive placebo in the double-blind feeder study AZES and switched to LY3314814 at the start of study AZFD did not "catch up" on the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog13) at Week 26 of study AZFD to participants originally randomized to receive LY3314814 in the double-blind feeder study.

ELIGIBILITY:
Inclusion Criteria:

* Participants previously enrolled in AMARANTH (NCT02245737) who meet eligibility criteria for delayed-start I8D-MC-AZFD.

Exclusion Criteria:

* Participants who participate in AMARANTH (NCT02245737) who develop new conditions precluding them from enrolling into I8D-MC-AZFD.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (132):
- United States (31):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Territory Neurology & Research Institute, Tucson, Arizona
  - Pacific Research Network Inc, San Diego, California
  - Mile High Research Center, Denver, Colorado
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Brain Matters Research, Delray Beach, Florida
  - Compass Research, Orlando, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Roskamp Institute, Sarasota, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - The Multiple Sclerosis Center of Atlanta, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Boston Center for Memory, Newton, Massachusetts
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - The Cognitive and Research Center of NJ, Springfield, New Jersey
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester School of Medicine, Rochester, New York
  - Valley Medical Primary Care, Centerville, Ohio
  - Lindner Research Center, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Radiant Research, Greer, South Carolina
  - Quillen College of Medicine, East TN State University, Johnson City, Tennessee
  - The Memory Clinic, Bennington, Vermont
- Australia (7):
  - Southern Neurology, Kogarah, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Eastern Clinical Research Unit, Box Hill, Victoria
  - Delmont Private Hospital, Glen Iris, Victoria
  - The Florey Institute of Neuroscience and Mental Health, Parkville, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia
  - Neuro Trials Victoria Pty Ltd, Noble Park
- Belgium (6):
  - Jessa Ziekenhuis, Hasselt, Limburg
  - Hopital Universitaire Brugmann Brussel, Brussels
  - Hospital Universitaire Erasme Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - AZ Delta, Roeselare
- Canada (9):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - True North Clinical Research Halifax, LLC, Halifax, Nova Scotia
  - Elizabeth Bruyere Health Centre, Ottawa, Ontario
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Clinique de la Memoire de l'Outaouais, Gatineau, Quebec
  - NeuroSearch Developements, Greenfield Park, Quebec
  - Hopital de L'Enfant Jesus, Québec, Quebec
  - Q&T Research Sherbrooke Inc, Sherbrooke, Quebec
- France (11):
  - Centre Hospitalier Universitaire La Timone, Marseille, Cedex 05
  - CHRU de Lille- Hôpital Roger Salengro, Lille, Cedex
  - CHU de Toulouse Hopital Purpan, Toulouse, Cedex
  - Hopital Neuro Pierre Wertheimer, Bron
  - CHU Bocage CMRR, Dijon
  - Hopital Broca, Paris
  - Hôpital de la Pitié-Salpêtrière, Paris
  - Hôpital Fernand Widal, Paris
  - Chu de Nantes Hopital Laennec, Saint-Herblain
  - Centre de Recherche Clinique du Gérontopôle Cité de la Santé, Toulouse
  - Hopital des Charpennes, Villeurbanne
- Germany (9):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Studien und Gedächtniszentrum München, München, Bavaria
  - Klinikum Rechts der Isar der TU München, München, Bavaria
  - Gemeinschaftspraxis für Neurologie und Psychiatrie, Westerstede, Lower Saxony
  - DataMed Klinische Studien GmbH, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Neurologische Praxis Siegen, Siegen, North Rhine-Westphalia
  - Pharm Studienzentrum Chemnitz, Mittweida, Saxony
  - Charité Universitätsmedizin Berlin, Berlin
- SE Neurologiai Klinika, Budapest, Hungary
- Japan (18):
  - National Institute for Longevity Sciences NCGG, Ōbu, Aichi-ken
  - National Chiba-East-Hospital, Chuo-ku, Chiba
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Iwate Medical University Hospital, Morioka, Iwate
  - Nihon Kokan Hospital, Kawasaki, Kanagawa
  - Katayama Medical Clinic, Kurashiki, Okayama-ken
  - Shiroma Clinic, Urasoe, Okinawa
  - Sakaguchi Clinic, Sakai, Osaka
  - National Sanatorium Toneyama Hospital, Toyonaka, Osaka
  - Memory Clinic Ochanomizu, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital, Bunkyo-Ku, Tokyo
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - National Sanatorium Hokuriku Hospital, Nanto, Toyama
  - Fukuoka University Hospital, Fukuoka
  - Kyoto University Hospital, Kyoto
  - Utano Hospital, Kyoto
  - Osaka City University Hospital, Osaka
- Poland (8):
  - Podlaskie Centrum Psychogeriatrii, Bialystok, Podlaskie Voivodeship
  - NZOZ Dom Sue Ryder - Pallmed Sp. z o.o., Bydgoszcz
  - NZOZ Wielospecjalistyczna Poradnia Lekarska, Katowice
  - Centrum Zdrowia Psychicznego Biomed - Jan Latala, Kielce
  - Krakowska Akademia Neurologii, Krakow
  - Medycyna Milorzab, Lodz
  - Instytut Medycyny Wsi, Lublin
  - Centrum Medyczne Neuroprotect, Warsaw
- Santa Cruz Behavioral PSC, Bayamón, Puerto Rico
- Romania (2):
  - SC Med Life SA, Bucharest
  - SC Centrul Medical Sana SRL, Bucharest
- South Korea (7):
  - Dong-A University Medical Center, Seogu, Busan
  - Hanyang University Guri Hospital, Guri-si, Gyeonggido
  - Inha University Hospital, Junggu, Incheon
  - Samsung Medical Center, Seoul, Korea
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
- Spain (14):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Virgen Del Puerto, Plasencia, Caceres
  - Hospital Universitario De Getafe, Madrid, Getafe
  - CITA Alzheimer, Donostia / San Sebastian, Guipuzcoa
  - Centro de Atencion Especializada (CAE) OROITU, Getxo, Vizcaya
  - Fundacion ACE-Institut Catala de Neurociences Aplicades, Barcelona
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital De La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Universitario Dr Pesset, Valencia
  - Hospital Universitario La Fe de Valencia, Valencia
- United Kingdom (8):
  - Re-Cognition Health Ltd, London, Greater London
  - MAC Clinical Research-Manchester, Manchester, Greater Manchester
  - MAC Clinical Research, Blackpool, Lancashire
  - West London Mental Health NHS Trust, Isleworth, London
  - MAC Clinical Research, Cannock, Staffordshire
  - Re-Cognition Health Ltd, Guildford, Surrey
  - Glasgow Memory Clinic, Glasgow
  - MAC Clinical Research, Leeds

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- See also: Click here for more information about this study: A Study of LY3314814 in Early Alzheimer's Disease Dementia — https://www.lillytrialguide.com/en-US/studies/alzheimer-s/AZFD#?postal=
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=16557&attachmentIdentifier=a046bc93-718a-4179-8f30-4b65da56a317&fileName=CSP_NCT02972658.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=16557&attachmentIdentifier=a6ee5d0a-4796-4efd-b082-e84fbcbac489&fileName=SAP_NCT02972658.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed feeder study [AZES (NCT02245737)] were enrolled in this study.
Pre-assignment Details: Participants who were randomized in Study AZES to either 20 milligrams (mg) or 50 mg of lanabecestat continued on the treatment allocation from the feeder study. Participants randomized to placebo in Study AZES were randomized in a blinded fashion, 1:1 ratio, to either lanabecestat 20 mg or 50 mg daily (QD), administered orally.
Groups:
- AZES Lanabecestat 20 mg/AZFD Lanabecestat 20 mg: Participants who received Lanabecestat 20 mg in the feeder study (AZES) were randomized to receive Lanabecestat 20 mg.
Period: Overall Study
Arm/Group | AZES Placebo/AZFD Lanabecestat 20 mg | AZES Lanabecestat 20 mg/AZFD Lanabecestat 20 mg | AZES Placebo/AZFD Lanabecestat 50 mg | AZES Lanabecestat 50 mg/AZFD Lanabecestat 50 mg
Started | 76 | 139 | 75 | 131
Received at Least 1 Dose of Study Drug | 76 | 139 | 74 | 131
Completed | 0 | 1 (1 participant was incorrectly marked as "Completed" rather than study terminated by Sponsor.) | 0 | 0
Not Completed | 76 | 138 | 75 | 131
Not completed — Adverse Event | 0 | 3 | 0 | 2
Not completed — Other-determined by Investigator | 1 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 2
Not completed — Progressive Disease | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 4 | 1 | 6
Not completed — Withdrawal due to Caregiver Circumstance | 1 | 1 | 1 | 0
Not completed — Sponsor Decision | 70 | 127 | 72 | 119

BASELINE CHARACTERISTICS:
Population: All randomized participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZES Placebo/AZFD Lanabecestat 20 mg | AZES Lanabecestat 20 mg/AZFD Lanabecestat 20 mg | AZES Placebo/AZFD Lanabecestat 50 mg | AZES Lanabecestat 50 mg/AZFD Lanabecestat 50 mg | Total
Number analyzed (Participants) | 76 | 139 | 75 | 131 | 421
Age, Continuous [Mean (Standard Deviation); unit: Years] — Details are from AZES baseline.
  Years | 70.7 (6.6) | 69.8 (7.8) | 71.1 (6.6) | 70.1 (6.7) | 70.3 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 76 | 40 | 75 | 226
  Male | 41 | 63 | 35 | 56 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 4 | 3 | 18
  Not Hispanic or Latino | 62 | 115 | 54 | 114 | 345
  Unknown or Not Reported | 7 | 20 | 17 | 14 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 7 | 23 | 10 | 16 | 56
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 0 | 3
  White | 64 | 104 | 51 | 106 | 325
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 10 | 13 | 9 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 0 | 1 | 0 | 0 | 1
  Romania | 1 | 1 | 0 | 0 | 2
  Hungary | 1 | 0 | 0 | 0 | 1
  United States | 23 | 35 | 13 | 23 | 94
  Japan | 6 | 14 | 5 | 14 | 39
  United Kingdom | 8 | 17 | 8 | 13 | 46
  Spain | 10 | 21 | 8 | 21 | 60
  Canada | 6 | 8 | 5 | 14 | 33
  South Korea | 1 | 7 | 3 | 2 | 13
  Belgium | 5 | 2 | 0 | 4 | 11
  Poland | 6 | 8 | 6 | 14 | 34
  France | 4 | 9 | 12 | 8 | 33
  Australia | 3 | 13 | 8 | 6 | 30
  Germany | 2 | 3 | 7 | 12 | 24
ADAS-Cog13 (13-item Alzheimer's Disease Assessment Scale) [Mean (Standard Deviation); unit: Units on a Scale] — ADAS-Cog13, a 13-item rating scale, measured the severity of cognitive dysfunction in persons with Alzheimer's disease (AD). Scores ranged from 0 to 85, with a higher score indicating worse cognitive functioning. Details are from AZES baseline.
  Units on a Scale | 27.9 (8.3) | 29.6 (7.8) | 27.0 (7.5) | 27.1 (7.5) | 27.9 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Analysis on the 13-item Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13)
Description: ADAS-Cog13 (13-item version of ADAS-Cog) is a psychometric instrument that evaluates word recall, ability to follow commands, constructional praxis, naming, ideational praxis, orientation, word recognition, memory, comprehension of spoken language, word-finding, and language ability, with a measure of delayed word recall and concentration/ distractibility. The total score of the 13-item scale ranges from 0 to 85, with an increase in score indicating cognitive worsening. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with factors for treatment, visit, treatment*visit, baseline efficacy score, baseline efficacy score-by-visit interaction, disease status at baseline, apolipoprotein E4 (APOE4) status, acetylcholinesterase inhibitor (AChEI) use at baseline, age at baseline, and pooled country.
Time Frame: AZES Baseline through AZFD Week 26
Population: All AZFD participants who received at least one dose of study drug and have baseline and at least one post-baseline data for ADAS-Cog13 measure. Feeder study AZES was stopped for futility, the original Delayed Start analysis was replaced with MMRM analysis and no comparisons between treatment groups were made.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- AZES Placebo/AZFD Lanabecestat 20 mg: Participants who received placebo in the feeder study (AZES) received Lanabecestat 20 mg in AZFD.
- AZES Lanabecestat 20 mg/AZFD Lanabecestat 20 mg: Participants who received Lanabecestat 20 mg in the feeder study (AZES) received Lanabecestat 20 mg in AZFD.
- AZES Placebo/AZFD Lanabecestat 50 mg: Participants who received placebo in the feeder study (AZES) received Lanabecestat 50 mg in AZFD.
- AZES Lanabecestat 50 mg/AZFD Lanabecestat 50 mg: Participants who received Lanabecestat 50 mg in the feeder study (AZES) received Lanabecestat 50 mg in AZFD.
Arm/Group | AZES Placebo/AZFD Lanabecestat 20 mg | AZES Lanabecestat 20 mg/AZFD Lanabecestat 20 mg | AZES Placebo/AZFD Lanabecestat 50 mg | AZES Lanabecestat 50 mg/AZFD Lanabecestat 50 mg
Number analyzed (Participants) | 76 | 139 | 75 | 131
Units on a scale | 9.61 (1.60) | 9.25 (1.21) | 8.41 (1.65) | 10.41 (1.25)

2. Secondary Outcome: Change From Baseline Analysis on the Alzheimer´s Disease Cooperative Study Activities of Daily Living Inventory Instrumental Items (ADCS-iADL)
Description: The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The ADCS-ADL measures both basic and instrumental activities of daily living by participants. The range for the ADCS-iADL is 0-59 with higher scores reflecting better performance. LS Mean was determined by MMRM with factors for treatment, visit, treatment*visit, baseline efficacy score, baseline efficacy score-by-visit interaction, disease status at baseline, APOE4 status, AChEI use at baseline, age at baseline, and pooled country.
Time Frame: AZES Baseline through AZFD Week 26
Population: All AZFD participants who received at least one dose of study drug and have baseline and at least one post-baseline data for ADCS-iADL measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZES Placebo/AZFD Lanabecestat 20 mg | AZES Lanabecestat 20 mg/AZFD Lanabecestat 20 mg | AZES Placebo/AZFD Lanabecestat 50 mg | AZES Lanabecestat 50 mg/AZFD Lanabecestat 50 mg
Number analyzed (Participants) | 76 | 139 | 74 | 129
Units on a scale | -9.19 (1.47) | -8.45 (1.10) | -7.37 (1.51) | -7.48 (1.14)

3. Secondary Outcome: Change From Baseline on the Functional Activities Questionnaire (FAQ) Score
Description: FAQ is a 10-item, caregiver-questionnaire and was administered to the study partner and asked to rate the participant's ability to perform a variety of activities ranging from writing checks, assembling tax records, shopping, playing games, food preparation, traveling, keeping appointments, traveling out of neighborhood, keeping track of current events and understanding media. FAQ total score was calculated by adding the scores from each of the 10 items. Each activity is rated on a scale from 0 to 3 (Never did and would have difficulty now =1; Never did but could do now =0; Normal =0; Has difficulty but does by self =1; Requires assistance =2; Dependent =3). FAQ scale is 0 to 30, with higher scores indicating greater impairment. LS Mean was determined by MMRM with factors for treatment, visit, treatment*visit, baseline efficacy score, baseline efficacy score-by-visit interaction, disease status at baseline, APOE4 status, AChEI use at baseline, age at baseline, and pooled country.
Time Frame: AZES Baseline through AZFD Week 26
Population: All AZFD participants who received at least one dose of study drug and have baseline and at least one post-baseline data for FAQ score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZES Placebo/AZFD Lanabecestat 20 mg | AZES Lanabecestat 20 mg/AZFD Lanabecestat 20 mg | AZES Placebo/AZFD Lanabecestat 50 mg | AZES Lanabecestat 50 mg/AZFD Lanabecestat 50 mg
Number analyzed (Participants) | 76 | 137 | 74 | 130
Units on a scale | 6.28 (0.98) | 7.09 (0.76) | 6.73 (1.01) | 6.91 (0.79)

4. Secondary Outcome: Change From Baseline on the Integrated Alzheimer's Disease Rating Scale (iADRS) Score
Description: The iADRS is a composite that measures both cognition and function. The iADRS comprises scores form the ADAS- Cog and the ADCS-iADL. The iADRS is calculated as a linear combination of the total scores of the ADAS-Cog13 (score range 0 to 85 with higher scores reflecting worse performance) and the ADCS-iADL (score range from 0-59 with higher scores reflecting better performance). The iADRS score ranges from 0 to 144 with higher scores indicating greater impairment. LS Mean was determined by MMRM with factors for treatment, visit, treatment*visit, baseline efficacy score, baseline efficacy score-by-visit interaction, disease status at baseline, APOE4 status, AChEI use at baseline, age at baseline, and pooled country.
Time Frame: AZES Baseline through AZFD Week 26
Population: All AZFD participants who received at least one dose of study drug and have baseline and at least one post-baseline data for iADRS.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZES Placebo/AZFD Lanabecestat 20 mg | AZES Lanabecestat 20 mg/AZFD Lanabecestat 20 mg | AZES Placebo/AZFD Lanabecestat 50 mg | AZES Lanabecestat 50 mg/AZFD Lanabecestat 50 mg
Number analyzed (Participants) | 76 | 138 | 72 | 123
Units on a scale | -18.85 (2.58) | -17.57 (1.97) | -15.37 (2.76) | -18.37 (2.09)

5. Secondary Outcome: Change From Baseline on the Mini-Mental Status Examination (MMSE)
Description: The MMSE is an instrument used to assess a participant's cognitive function. The MMSE assesses orientation to time and place, immediate and delayed recall of words, attention and calculation, language (naming, comprehension and repetition), and spatial ability (copying a figure). The range for MMSE total Score is 0 to 30, with a higher score indicating better cognitive performance. LS Mean was determined by MMRM methodology with factors for treatment, visit, treatment*visit, baseline efficacy score, baseline efficacy score-by-visit interaction, disease status at baseline, APOE4 status, AChEI use at baseline, age at baseline, and pooled country.
Time Frame: AZES Baseline through AZFD Week 26
Population: All AZFD participants who received at least one dose of study drug and have baseline and at least one post-baseline data for MMSE.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZES Placebo/AZFD Lanabecestat 20 mg | AZES Lanabecestat 20 mg/AZFD Lanabecestat 20 mg | AZES Placebo/AZFD Lanabecestat 50 mg | AZES Lanabecestat 50 mg/AZFD Lanabecestat 50 mg
Number analyzed (Participants) | 76 | 139 | 75 | 131
Units on a scale | -5.84 (0.71) | -5.73 (0.54) | -4.72 (0.72) | -5.25 (0.56)

6. Secondary Outcome: Change From Baseline Analysis on the ADAS-Cog13
Description: ADAS-cog13 (13-item ADAS cog) is a psychometric instrument that evaluates word recall, ability to follow commands, constructional praxis, naming, ideational praxis, orientation, word recognition, memory, comprehension of spoken language, word-finding, and language ability, with a measure of delayed word recall and concentration/ distractibility. The total score of the 13-item scale ranges from 0 to 85, with an increase in score indicating cognitive worsening. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with factors for treatment, visit, treatment*visit, baseline efficacy score, baseline efficacy score-by-visit interaction, disease status at baseline, APOE4 status, AChEI use at baseline, age at baseline, and pooled country.
Time Frame: AZES Baseline through AZFD Week 52
Population: All AZFD participants who received at least one dose of study drug and have baseline and at least one post-baseline data for ADAS-Cog13 measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZES Placebo/AZFD Lanabecestat 20 mg | AZES Lanabecestat 20 mg/AZFD Lanabecestat 20 mg | AZES Placebo/AZFD Lanabecestat 50 mg | AZES Lanabecestat 50 mg/AZFD Lanabecestat 50 mg
Number analyzed (Participants) | 76 | 139 | 75 | 131
Units on a scale | 16.64 (3.45) | 12.40 (2.25) | 16.79 (2.47) | 15.05 (2.06)

ADVERSE EVENTS:
Time Frame: Up To 156 Weeks
Description: All AZFD participants who received at least one dose of study drug.
Arm/Group | AZES Placebo/AZFD Lanabecestat 20 mg | AZES Lanabecestat 20 mg/AZFD Lanabecestat 20 mg | AZES Placebo/AZFD Lanabecestat 50 mg | AZES Lanabecestat 50 mg/AZFD Lanabecestat 50 mg
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/139 | 0/74 | 1/131
Serious Adverse Events (participants affected / at risk) | 3/76 | 8/139 | 5/74 | 7/131
Other Adverse Events (participants affected / at risk) | 11/76 | 23/139 | 8/74 | 17/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZES Placebo/AZFD Lanabecestat 20 mg (N=76) | AZES Lanabecestat 20 mg/AZFD Lanabecestat 20 mg (N=139) | AZES Placebo/AZFD Lanabecestat 50 mg (N=74) | AZES Lanabecestat 50 mg/AZFD Lanabecestat 50 mg (N=131)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiation proctitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram repolarisation abnormality (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropsychiatric symptoms (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZES Placebo/AZFD Lanabecestat 20 mg (N=76) | AZES Lanabecestat 20 mg/AZFD Lanabecestat 20 mg (N=139) | AZES Placebo/AZFD Lanabecestat 50 mg (N=74) | AZES Lanabecestat 50 mg/AZFD Lanabecestat 50 mg (N=131)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 8 (8) | 2 (2) | 6 (6)
Nasopharyngitis (Infections and infestations) | 1 (1) | 8 (10) | 3 (3) | 5 (7)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 7 (8) | 3 (3) | 5 (8)
Depression (Psychiatric disorders) | 4 (4) | 3 (3) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
This study was stopped after an independent assessment concluded that the feeder study AZES was futile. Because of this, the originally planned delayed-start analysis for this study was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor shall review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. Investigator shall delay publication of their results of the study until the results of the multi-center study are published or presented, provided the multi-center results are published within 24 months of the termination.

DOCUMENTS (2):
  • Study Protocol (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT02972658/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT02972658/SAP_001.pdf